CLINICAL TRIAL: NCT00261690
Title: Use of Virtual Reality for Adjunctive Treatment of Burn Pain
Brief Title: Virtual Reality Pain Control During Burn Wound Care
Acronym: VRPT/H2O/RT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David R. Patterson, PhD, ABPP. Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13289-C; R01GM042725 (NIH)
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2012-06

CONDITIONS: Burn
Keywords: Virtual Reality Distraction
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Virtual Reality distraction
  Interventions: Behavioral: Virtual Reality Distraction

INTERVENTIONS:
Behavioral: Virtual Reality Distraction — Using virtual reality distraction during a procedure

SUMMARY:
Using Virtual Reality as a form of Distraction during Burn Care.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effectiveness of virtual reality (a form of distraction) in order to reduce patients' procedural burn pain.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete subjective evaluations of pain
* English-speaking
* Not demonstrating delirium, psychosis, or any form of Organic Brain Disorder
* Able to communicate orally

Exclusion Criteria:

* Incapable of indicating subjective evaluation of pain
* Non-English-speaking
* Severe head or neck injury or other medical conditions that prohibit patient from wearing VR helmet
* Demonstrating delirium, psychosis, or Organic Brain Disorder
* Unable to communicate verbally
* Significant developmental disability
* Extreme susceptibility to motion sickness
* Reports having no problem with pain during wound care.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2002-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
We use GRS, McGill to measure the outcome. | once a day

CONTACTS AND LOCATIONS:
Overall Officials: David R. Patterson, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington; Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Hoffman HG, Patterson DR, Magula J, Carrougher GJ, Zeltzer K, Dagadakis S, Sharar SR. Water-friendly virtual reality pain control during wound care. J Clin Psychol. 2004 Feb;60(2):189-95. doi: 10.1002/jclp.10244. PMID 14724926